CLINICAL TRIAL: NCT04449107
Title: To Evaluate the Role of a Personalized Smartphone-based Application to Improve Childhood Immunization Coverage and Timelines Among Children in Pakistan
Brief Title: Evaluate the Role of a Personalized Smartphone Based Application to Improve Childhood Immunization Coverage
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Aga Khan University (Other)
Collaborators: NED University of Engineering and Technology (Unknown); University of Surrey (Other)
Responsible Party: Principal Investigator, Dr Abdul Momin Kazi, Assistant Professor, Aga Khan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2019-1534-5556
Record Dates: First submitted 2020-04-14; First posted 2020-06-26 (Actual); Last update posted 2020-06-26 (Actual); Status verified 2020-06

CONDITIONS: Mobile Application; Routine Childhood Immunization
Keywords: Mobile application; routine childhood immunization

STUDY DESIGN:
Intervention Model Description: A mixed methods study will be conducted in which a smart phone application will be developed based on the findings of qualitative component of the study, which will have features for text, voice, video and pictorial messages for the participant caregivers to improve RI on 10th and 14th week of child age.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Experimental): The intervention arm in addition to the standard counselling will include receiving text messages, voice messages, pictorial messages and video messages regarding vaccination once a week till the child turns 14 weeks
  Interventions: Behavioral: Android based mobile phone application
- Control Arm (No Intervention): The control group will receive one-time standard verbal counselling at the time of initial visit for on-time EPI vaccines at 10 and 14 weeks of age as recommended by EPI, government of Pakistan.

INTERVENTIONS:
Behavioral: Android based mobile phone application — An android based mobile application will be developed. The application will have features and capacity for text messages, voice messages, pictorial messages and video messages. The content of the messages will be according to the findings of Paigham e sehat project and the four messages domains would be educational, reminder, religious and adverse effects. In addition, pictorial and video messages would be used as per freely available through EPI programme Pakistan.
  Arms: Intervention Arm

SUMMARY:
The vision of the investigators is to build capacity in technology-driven healthcare innovation in LMCIs. The programme will be initiated by a feasibility and proof-of-concept (POC) study to tackle the lack of awareness around immunization, which is a major health issue in developing countries. Mobile apps and social media have been shown to be effective in various programmes worldwide, but there is limited data from LMICs on the use of digital technologies in improving routine immunization (RI) coverage.

DETAILED DESCRIPTION:
Pakistan is one of the countries with the highest rates of child death in the world. It ranks 4th in child mortality, with 60% deaths due to vaccine-preventable diseases (VPDs). The immunization coverage in Pakistan is estimated to be 59%, which is still well below the desired level, leading to continued polio transmission, large measles outbreaks, and thousands of deaths from vaccine-preventable illnesses. In addition, Pakistan is a major polio epidemic country and among 3 countries in the world requiring proof of polio vaccination for international travel. Pakistan demographic and health survey in 2017-2018 suggests 88% percent of children had received BCG vaccine due at birth, 86% and 95% had received the first dose of pentavalent and polio vaccine respectively due at the 6th week. Furthermore, 75% and 86% of children had received the third dose of the pentavalent and polio vaccines, respectively, due at 14th week and measles vaccination was 73%, which is due at 9 months. However, these rates are at 1 year of age and much higher than vaccination coverage rate at scheduled time and among conflict hits and displaced populations. Improved RI coverage is recommended as the priority public health strategy to reduce VPDs and eradicate polio in Pakistan and worldwide.

According to immunization coverage surveys, 1 in 5 children are unimmunized. A major reason for poor childhood vaccine coverage is low immunization uptake, when parents are unable to complete the entire series of vaccines in accordance with the scheduled timelines. Some of the reasons include: (1) the family is not in favor of getting their child immunized, (2) low trust in vaccines provided through Expanded Programme on Immunization (EPI) and government health care providers, and (3) caregivers have forgotten their child's next vaccination due date or child's EPI card is misplaced. These barriers may be modified with additional support through education and behavior change strategies. In addition, with more pressing issues of food and shelter, preventive health often takes the back seat, and parents and caregivers forget or ignore the subsequent doses of vaccines for their children. There is an immense need to encourage parents' care seeking and collaboration with the health care providers to improve initial vaccine uptake and the completion of all doses according to the schedule. New innovative and cost-effective techniques are necessary for practical solutions to improve vaccination uptake and coverage.

Mobile phones offer a new medium to provide education and advocate families or caregivers to enable behavior change so as to improve immunization uptake. Mobile phone use has also increased in countries with low RI coverage and a high risk of VPDs. Good examples are Nigeria and Pakistan, where there were around 170 and 140 million mobile phone subscribers, respectively, in 2014. There are limited data from LMICs set up on the role of SMS-based interventions for improvement of RI coverage, and conventional 1-way reminder SMS text messages were used by most of the studies as the intervention. Overall, very few studies compared reminders, educational, and interactive SMS messages related to childhood vaccination uptake. Although some of the studies have shown some behavior change for improvement in vaccination coverage, more rigorous application of health behavior change model needs to be applied to understand the impact of reminder, educational, and interactive messages on behavior change related to improvement in RI coverage. However, data from developing countries regarding the role of automated calls in improving vaccine coverage are limited.

The vision of the investigators is to build capacity in technology-driven healthcare innovation in LMCIs. The programme will be initiated by a feasibility and proof-of-concept (POC) study to tackle the lack of awareness around immunization, which is a major health issue in developing countries. Mobile apps and social media have been shown to be effective in various programmes worldwide, but there is limited data from LMICs on the use of digital technologies in improving routine immunization (RI) coverage.

ELIGIBILITY:
Inclusion Criteria:

* parent or guardian or at least one person in the household has a working android based smart mobile phone
* ability to use android based smart phone
* Parent or guardian providing consent.

Exclusion Criteria:

* If the family will not be visiting AKU for 10- and 14-week RI.

Ages: 6 Weeks to 2 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 328 (Actual)
Dates: Start 2020-02-27 (Actual); Primary Completion 2020-08-30 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
improvement in RI coverage | 12 weeks
  to see a 10 percent increase in RI through personalized smart mobile phone-based application at 10 and 14 weeks of age according to the EPI schedule versus standard care
Improvement in timeline | 12 weeks
  To see a 10 percent increase in RI within 1 week of the original timeline at 10, and 14 weeks versus standard care

SECONDARY OUTCOMES:
Perceptions and barriers related to routine immunization (Interview guide in form of in depth interview will be administered). | 6 weeks
  1. Perceptions regarding risks of infectious diseases preventable by vaccines and vaccine safety and efficacy.
  2. Perceptions and barriers to vaccinating children including difficulties in visiting RI centers.
  This will help us in understanding the types of (1) barriers perceived by caregivers, (2) designing the Randomized Controlled Trial and study methodology.
perceptions and barriers of a mobile phone based application to improve immunization coverage (interview guide in form of in depth interview will be administered) | 4 weeks
  1. Perceptions and barriers that may affect the use of mobile phone application in implementing the phone-based intervention to improve immunization coverage
  2. Usability and preferences of mobile phone app to improve routine immunization coverage
  This will help in developing personalized mobile phone application and content of the messages according to the barriers of the participants to bring in behavior change in order to improve immunization coverage and timelines
  Measurement tool is the 14 weeks vaccination as per EPI schedule.

CONTACTS AND LOCATIONS:
Locations (1):
- Aga Khan University, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No
The database will reside on a central computer at AKU managed by the study staff. Mobile numbers will not be shared except to track patterns of use. Only relevant study staff will have access to study data allowed by the local ethics committee. Participants' information will be given a study code, and no personal identifiers will be shared. Data confidentiality will be maintained at all times. No personal identifiers will be used in any reports or publication of the study. No individual identifier such as names of participants and area of location will be shared. In addition, a confidentiality agreement has been signed with the universities stating that the numbers provided will only be used for the purpose of the trial.

REFERENCES:
- [Derived] Kazi AM, Qazi SA, Khawaja S, Ahsan N, Ahmed RM, Sameen F, Khan Mughal MA, Saqib M, Ali S, Kaleemuddin H, Rauf Y, Raza M, Jamal S, Abbasi M, Stergioulas LK. An Artificial Intelligence-Based, Personalized Smartphone App to Improve Childhood Immunization Coverage and Timelines Among Children in Pakistan: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2020 Dec 4;9(12):e22996. doi: 10.2196/22996. PMID 33274726